## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | Ī | Reporting and Analysis Plan for Study BTZ117351: A Phase I, Multi-Center, Open-Label (Parts 1 and 2); Randomized, Double-Blind, Placebo-Controlled (Part 3); Single-Dose; 3-Part Study to Evaluate the Relative Bioavailability of Three Formulations in Healthy Subjects, Food Effect on Tablet Formulation in Healthy Subjects, and Pharmacokinetics of Gepotidacin (GSK2140944) in Japanese Subjects in Fasted and Fed States |
|---|---|---|
| <b>Compound Number</b> | : | GSK2140944 |
| Effective Date | : | 27-NOV-2017 |

## **Description:**

- This RAP is amended from the original version dated 05-OCT-2016. The RAP has been updated per the changes from Protocol Amendment 2.
- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol BTZ117351.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | Ph.D. | 27-NOV-2017 |
|---|---|---|
| Biostatisticia | Biostatistician II (Biostatistics, Early Development Services, PPD) | |
| PPD | Pharm.D. | 27-NOV-2017 |
| Pharmacokin | eticist (Biostatistics, Phase II-IV, PPD) | 2/-INOV-201/ |

## Approved by:

| PPD | Ph.D. | 27-NOV-2017 |
|---|---|---|
| Director Clinical Statis | Director Clinical Statistics, GSK | |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN S | SYNOPSIS | 4 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | Changes<br>Study O<br>Study De | to the Protocol De<br>jective(s) and End<br>sign | NFORMATIONfined Statistical Analysis Planpoint(s) | 7<br>7 |
| 3. | PLANI<br>3.1.<br>3.2. | Interim A | nalyses | | <mark>11</mark> |
| 4. | ANAL`<br>4.1. | | | | |
| 5. | | | | NALYSES AND DATA HANDLING | 13 |
| 6. | STUD<br>6.1. | | | ses | |
| 7. | PRIMA<br>7.1. | | okinetic Analyses Overview of Plann Drug Concentratio Pharmacokinetic F 7.1.3.1. Derivin 7.1.3.2. Statistic Paramo Interim Analysis | ed Pharmacokinetic Analyses | |
| 8. | SECO<br>8.1. | | | YSES | |
| 9. | REFE | RENCES | | | 24 |
| 10. | APPE<br>10.1.<br>10.2. | Appendi<br>10.1.1. | 1: Time & Events. Protocol Defined 1 | Fime & Eventses and Phases | 26 |
| | 10.2. | 10.2.1. | Treatment States 10.2.1.1. Treatm 10.2.1.2. Treatm | ent States for Safety Dataent States for AE Data | 28<br>28<br>28 |
| | 10.3. | Appendi<br>10.3.1.<br>10.3.2. | Study Treatment & Baseline Definition | tandards & Handling Conventions<br>& Sub-group Display Descriptors<br>n & Derivations<br>ne Definitions | 29<br>29 |

| | | 10.3.2.2. | Derivations and Handling of Missing Baseline | |
|---|---|---|---|---|
| | | | Data | 30 |
| | 10.3.3. | Reporting | Process & Standards | 30 |
| 10.4. | Appendix | 4: Derived | I and Transformed Data | 33 |
| | 10.4.1. | General | | 33 |
| | 10.4.2. | Study Pop | ulation | 33 |
| | 10.4.3. | Safety | | 3 <mark>3</mark> |
| 10.5. | Appendix | 5: Premat | ure Withdrawals & Handling of Missing Data | 35 |
| | 10.5.1. | Premature | Withdrawals | 35 |
| | 10.5.2. | | of Missing Data | |
| | | 10.5.2.1. | Handling of Missing Dates | 35 |
| | | 10.5.2.2. | Handling of Partial Dates | 36 |
| 10.6. | | | of Potential Clinical Importance | |
| | | | 3 | 37 |
| 10.7. | | | n of Microbiology and Infectious Disease Adult | |
| | | | Adverse Event Assessment | |
| | | | / Values | |
| 10.8. | | | Comparisons & Multiplicity | |
| | | | of Multiple Comparisons & Multiplicity | 41 |
| 10.9. | | | Checking and Diagnostics for Statistical | |
| | | | Analysis Assumptions | |
| 10.10. | | | eviations & Trade Marks | |
| | | | ons | |
| | | | (S | |
| 10.11. | | | Data Displays | |
| | | | ay Numbering | |
| | | | mple Referencing | |
| | | | e [Priority] | |
| | | , , | ulation Tables | |
| | | | bles | |
| | | | kinetic Tables | |
| | | | kinetic Figures | |
| | 10.11.8. | ICH Listing | gs | 53 |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | <ul> <li>The purpose of this reporting and analysis plan (RAP) is to describe any planned<br/>analyses and output to be included in the clinical study report for Protocol<br/>BTZ117351.</li> </ul> |
| Protocol | This RAP is based on protocol amendment 2 (Dated: 05-SEP-2017) for study BTZ117351 [GlaxoSmithKline Document Number: 2016N281831_02. |
| Primary | Part 1a: |
| Objective | <ul> <li>Evaluate the relative bioavailability of a single 1500 mg dose of gepotidacin free<br/>base tablet formulations (related compound (RC) and high shear wet granulation<br/>(HSWG); 2 × 750 g) compared to the reference capsule formulation<br/>(3 × 500 mg).</li> </ul> |
| | Part 1b: |
| | <ul> <li>Evaluate the effect of a moderate fat meal on the bioavailability of a single 1500<br/>mg (2 × 750 mg) dose of gepotidacin tablets (RC or HSWG) selected from<br/>Part 1a</li> </ul> |
| | Part 2: |
| | <ul> <li>Evaluate the pharmacokinetics of a single 1500 mg (2 × 750 mg) dose followed<br/>by a single 3000-mg (4 x 750 mg) does of gepotidacin tablets (RC or HSWG)<br/>selected from Part 1a in Japanese subjects</li> </ul> |
| | Part 3: |
| | <ul> <li>Evaluate the pharmacokinetics of a single 1500 mg (2 × 750 mg) dose, a single 2250 mg (3 × 750 mg) dose, and a single 3000 mg (4 × 750 mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects in the fed state</li> </ul> |
| Primary | Parts 1a, 2 and 3: |
| Endpoint | <ul> <li>Plasma gepotidacin AUC(0-∞), AUC(0-t), Frel (for Part 1a only), Cmax, tmax,<br/>tlag, and t1/2, as data permit.</li> </ul> |
| | <ul> <li>Urine endpoints include Ae total, Ae(t1-t2), AUC(0-12), AUC(0-24), AUC(0-48),<br/>fe%, and CLr of gepotidacin, as data permit.</li> </ul> |
| | Part 1b: |
| | <ul> <li>Plasma gepotidacin AUC(0-∞), AUC(0-t), Cmax, tmax, tlag, and t1/2, as data<br/>permit.</li> </ul> |
| Secondary | Part 1a: |
| Objective | <ul> <li>To assess the safety and tolerability of a single 1500 mg dose of gepotidacin<br/>tablet formulations (RC and HSWG; 2 × 750 mg) compared to the reference<br/>capsule formulation (3 × 500 mg)</li> </ul> |
| | Part 1b: |
| | <ul> <li>To assess the safety and tolerability of a single 1500 mg (2 × 750 mg) dose of<br/>gepotidacin tablets (RC or HSWG) selected from Part 1a when administered<br/>with a moderate fat meal</li> </ul> |
| | Part 2: |
| | To assess the safety and tolerability of a single 1500 mg (2 × 750 mg) dose |

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| | followed by a single 3000 mg (4 x 750 mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects |
| | <ul> <li>To assess dose proportionality following a single 1500 mg (2 × 750 mg) dose<br/>followed by a single 3000 mg (4 x 750 mg) dose of gepotidacin tablets (RC or<br/>HSWG) selected from Part 1a in Japanese subjects</li> </ul> |
| | Part 3: |
| | <ul> <li>To assess the safety and tolerability of a single 1500 mg (2 × 750 mg) dose, a<br/>single 2250 mg (3 × 750 mg) dose, and a single 3000 mg (4 × 750 mg) dose of<br/>gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects in<br/>the fed state</li> </ul> |
| | <ul> <li>To assess dose proportionality of a single 1500 mg (2 × 750 mg) dose, a single<br/>2250 mg (3 × 750 mg) dose, and a single 3000 mg (4 × 750 mg) dose of<br/>gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects in<br/>the fed state</li> </ul> |
| Secondary<br>Endpoint | Clinical safety data from adverse events (AEs), clinical laboratory tests, vital signs (systolic and diastolic blood pressure and heart rate), and 12-lead electrocardiogram (ECG) readings. |
| | <ul> <li>Plasma gepotidacin AUC(0-∞) and Cmax, as data permit (for Parts 2 and 3 only)</li> </ul> |
| Study<br>Design | • This is a Phase I, multi-center, open-label, single-dose, 3-part study. Part 1a is being conducted to evaluate the relative bioavailability of 2 free base tablet formulations of gepotidacin compared to the reference capsule formulation under fasted conditions. Based upon safety and pharmacokinetic (PK) data obtained from Part 1a, a decision will be made whether to use the free base RC or HSWG tablet formulation for Parts 1b and 2. Part 1b will evaluate the bioavailability of the selected tablet formulation under fasted and fed conditions. Part 2 will evaluate pharmacokinetics of 2 different doses of the formulation selected from Part 1a in Japanese subjects under fasted conditions. Part 3 will evaluate pharmacokinetics of 3 single escalating doses of the selected tablet formulation in Japanese subjects in the fed state. |
| | <ul> <li>Part 1a is a 3-period, cross-over study that will assess the relative bioavailability of a single 1500-mg dose of gepotidacin in 2 free base tablet formulations (2 × 750 mg RC and HSWG tablets) compared with the reference capsule formulation of Gepotidacin (3 × 500-mg capsules) under fasted conditions. Each subject will receive all 3 treatments according to their assigned treatment sequence based on a Latin square design (ABC, CAB, or BCA).</li> </ul> |
| | <ul> <li>Part 1b is a 2-period, cross-over study and will evaluate the effect of food on the<br/>safety, tolerability, and pharmacokinetics of a single dose of 1500 mg<br/>gepotidacin tablet formulation (selected in Part 1a).</li> </ul> |
| | <ul> <li>Part 2 is a 2-period, fixed-sequence study and will evaluate the pharmacokinetics of a single dose of 1500 mg followed by a single dose of 3000 mg gepotidacin tablet formulation (RC or HSWG tablet) in a cohort of Japanese subjects under fasted conditions. A decision will be made whether to use the RC tablet formulation or the HSWG tablet formulation based upon the safety and PK data obtained from Part 1a.</li> </ul> |
| | Part 3 is a 3-period, randomized, double-blind, placebo-controlled, fixed- |

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| | sequence study and will evaluate the safety tolerability, and pharmacokinetics of single ascending doses of 1500 mg, 2250 mg, and 3000 mg gepotidacin formulation selected from Part 1a or placebo in a cohort of Japanese subjects in the fed state. |
| Analysis<br>Population | Safety Population (All subjects who receive at least one dose of study drug and have at least 1 postdose safety assessment). |
| | <ul> <li>PK Population (All subjects who received at least 1 dose of gepotidacin and<br/>have evaluable PK data for gepotidacin).</li> </ul> |
| | <ul> <li>PK Parameter Population (All subjects in the PK population for whom valid and<br/>evaluable PK parameters were derived. This population will be used in the<br/>assessment and characterization of PK parameters).</li> </ul> |
| Hypothesis | <ul> <li>A formal hypothesis will not be tested; however, an estimation approach will be<br/>taken to characterize the relative bioavailability of the gepotidacin RC and<br/>HSWG tablet formulations relative to the reference gepotidacin capsule<br/>formulation in healthy subjects (Part 1a), estimate the effect of food on the tablet<br/>formulation selected in Part 1a (Part 1b), and to evaluate the pharmacokinetics<br/>of the tablet formulation selected in Part 1a in Japanese subjects (Parts 2 and<br/>3).</li> </ul> |
| Planned<br>Analyses | Safety and PK data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There was one change to the originally planned statistical analysis specified in protocol amendment 2 [Dated:05/SEP/2017]. For the fed Japanese subjects (Part 3), dose proportionality will be evaluated using a power model, in addition to dose-normalized PK parameters in the pooled analysis with Part 2.

# 2.2. Study Objective(s) and Endpoint(s)

| Obje | ectives | Endpoints | |
|---|---|---|---|
| | | Primary Endpoints | |
| Part | | Part | |
| • | To evaluate the relative bioavailability of a single 1500-mg dose of gepotidacin free base tablet | • | Plasma gepotidacin AUC(0- $\infty$ ), AUC(0-t), Frel, Cmax, tmax, tlag and t1/2, as data permit. |
| | formulations (RC and HSWG; 2 × 750 mg) compared to the reference capsule formulation (3 × 500 mg) | • | Urine endpoints include Ae total, Ae(t1-t2), AUC(0-12), AUC(0-24), AUC(0-48), fe%, and CLr of gepotidacin, as data permit. |
| Part | 1b | Part | : 1b |
| • | the bioavailability of a single 1500-mg (2 $\times$ 750 mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a | | Plasma gepotidacin AUC(0- $\infty$ ), AUC(0-t), Cmax, tmax, tlag, and t1/2, as data permit. |
| Part | 2 | Part | 12 |
| • | To evaluate the pharmacokinetics of a single 1500-mg ( $2 \times 750$ mg) dose followed by a single 3000-mg ( $4 \times 750$ mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects | • | Plasma gepotidacin AUC(0- $\infty$ ), AUC(0-t), Cmax, tmax, tlag, and t1/2, as data permit. Urine endpoints include Ae total, Ae(t1-t2), AUC(0-12), AUC(0-24), AUC(0-48), fe%, and CLr of gepotidacin, as data permit. |
| Part | <b>-</b> | Part | |
| • | To evaluate the pharmacokinetics of a single 1500-mg (2 × 750 mg) dose, a single 2250-mg | • | Plasma gepotidacin AUC(0-∞), AUC(0-t), Cmax, tmax, tlag, and t1/2, as data permit. Urine endpoints include Ae total, Ae(t1-t2), AUC(0-12), AUC(0-24), AUC(0-48), fe%, and CLr of gepotidacin, as data permit. |
| Sec | ondary Objectives | Sec | ondary Endpoints |
| Part | | | is 1a |
| • | | • | Clinical safety data from adverse events (AEs), clinical laboratory tests, vital signs (systolic and diastolic blood pressure and heart rate), and 12-lead electrocardiogram (ECG) readings. |
| Part | 1b | Part | : 1b |
| • | 1500-mg (2 × 750 mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a when administered with a moderate fat meal | • | Clinical safety data from AEs, clinical laboratory tests, vital signs (systolic and diastolic blood pressure and heart rate), and 12-lead ECG readings. |
| Part | | Part | |
| • | To assess the safety and tolerability of a single 1500-mg ( $2 \times 750$ mg) dose followed by a single 3000-mg ( $4 \times 750$ mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects | • | Clinical safety data from AEs, clinical laboratory tests, vital signs (systolic and diastolic blood pressure and heart rate), and 12-lead ECG readings. Plasma gepotidacin AUC(0-t), AUC(0-∞) and Cmax, as data permit. |

| Obj | ectives | Endpoints |
|---|---|---|
| • | To assess dose proportionality following a single 1500-mg (2 × 750 mg) dose followed by a single 3000-mg (4 x 750 mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1 in Japanese subjects | |
| Par | 13 | Part 3 |
| • | To assess the safety and tolerability of a single 1500-mg ( $2 \times 750$ mg) dose, a single 2250-mg ( $3750$ mg) dose, and a single 3000-mg ( $4 \times 750$ mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects in the fed state | <ul> <li>Clinical safety data from AEs, clinical laboratory tests, vital signs (systolic and diastolic blood pressure and heart rate), and 12-lead ECG readings.</li> <li>Plasma gepotidacin AUC(0-t), AUC(0-∞) and Cmax, as data permit.</li> </ul> |
| • | To assess dose proportionality following a single 1500-mg ( $2 \times 750$ mg) dose, a single 2250-mg ( $3 \times 750$ mg) dose, and a single 3000-mg ( $4 \times 750$ mg) dose of gepotidacin tablets (RC or HSWG) selected from Part 1a in Japanese subjects in the fed state | |

# 2.3. Study Design

## **Overview of Study Design and Key Features**

## Part 1a Relative Bioavailability

| Treatment | | Follow-up | | | | | |
|---|---|---|---|---|---|---|---|
| Capsule<br>(reference) <sup>a</sup><br>RC and<br>HSWG<br>tablet <sup>b</sup> | Period<br>1 | Wash-out<br>At least 3<br>days | Period<br>2 | Wash-out<br>At least 3<br>days | Period<br>3 | Wash-out<br>At least 3<br>days | 5 to 7 days<br>after final<br>dose |
| Sequence 1 | | Α | | В | | С | |
| Sequence 2 | | С | Α | | В | | _ |
| Sequence 3 | | В | | С | | Α | |

HSWG = high shear wet granulation, RC = related compound

- a 1500 mg single dose given as  $3 \times 500 \text{ mg}$  capsules (Treatment A; reference formulation) under fasted conditions
- b 1500 mg single does given as  $2 \times 750 \text{ mg}$  RC (Treatment B) or HSWG (Treatment C) tablets under fasted conditions

## Part 1b (Optional) Food Effect

| Treatment | | Cross-over | | Follow-up |
|---|---|---|---|---|
| RC or HSWG tablet fasted <sup>a</sup> RC or HSWG tablet fed <sup>a</sup> | Period 1 | Wash-out<br>At least<br>3 days | Period 2 | 5 to 7 days after final dose |
| Sequence 4 | | D | Е | |
| Sequence 5 | Е | | D | |

HSWG = high shear wet granulation, RC = related compound

a 1500 mg single dose given as 2 × 750 mg tablets fasted (Treatment D) and fed (Treatment E) conditions

## **Overview of Study Design and Key Features**

#### Part 2 Pharmacokinetic

| Treatment | | Sequence | Follow-up | |
|---|---|---|---|---|
| RC or HSWG tablet fasted <sup>a</sup> | Period 1 | Wash-out<br>At least 3<br>days | Period 2 | 5 to 7 days after final dose |
| Sequence 6 | B or C | | F | |

HSWG = high shear wet granulation, RC = related compound

#### Part 3 Pharmacokinetic - Fed State

| Treatment | | , | Sequence | (EGH or III) | | Follow-up |
|---|---|---|---|---|---|---|
| Capsule<br>(reference) <sup>a</sup><br>RC and<br>HSWG<br>tablet <sup>b</sup> | Period<br>1 | Wash-out<br>At least 3<br>days | Period 2 | Wash-out<br>At least 3<br>days | Period 3 | 5 to 7 days<br>after final<br>dose |
| Sequence 7 | Е | or I | G | or l | H or I | |

HSWG = high shear wet granulation, RC = related compound

# Design Features

- Phase I, multi-centre, single-dose, 3-part study.
- Part 1a: Approximately 27 subjects in a 3-period, cross-over study that will assess the relative bioavailability of gepotidacin in 2 free base tablet formulations (2 × 750 mg related compound (RC) [Treatment B] and high shear wet granulation (HSWG) tablets [Treatment C]) compared with the reference capsule formulations of gepotidacin (3 × 500 mg capsules [Treatment A]) under fasted conditions. Each subject will receive all 3 treatments according to their assigned treatment sequence based on a Latin square design (ABC, CAB, or BCA). Each cohort will contain 9 subjects.
- Based upon safety and pharmacokinetic (PK) data obtained from Part 1a, a decision will be made whether to use the free base RC or HSWG tablet formulation for Parts 1b and 2
- Part 1b: Approximately 16 subjects in a 2-period, cross-over study that will
  evaluate the bioavailability of the selected tablet formulation under fasted and
  fed conditions. Each cohort will contain 8 subjects.
- Part 2: Approximately 10 Japanese subjects in a 2-period, fixed-sequence study that will evaluate the pharmacokinetics of a single dose of 1500 mg (2 x 750 mg) followed by a single dose of 3000 mg (4 x 750 mg) gepotidacin tablet formulation (RC or HSWG tablet) under fasted conditions.
- Part 3: Approximately 12 Japanese subjects stratified by gender, randomized to

a 1500 mg single dose given as 2 × 750-mg RC (Treatment B) or HSWG (Treatment C) tablets; 3000 mg single dose given as 4 x 750-mg RC or HSWG tablets (Treatment F), both under fasted conditions

a 1500 mg single dose given as  $2 \times 750$ -mg RC or HSWG (Treatment E) tablets – fed; 2250 mg single dose given as  $3 \times 750$ -mg RC or HSWG (Treatment G) tablets – fed; 3000 mg single dose given as  $4 \times 750$ -mg RC or HSWG (Treatment H) tablets – fed; or placebo (Treatment I) tablets - fed

## **Overview of Study Design and Key Features**

active or placebo in a 5:1 ratio in a 3-period, double-blind, placebo-controlled, fixed-sequence study that will evaluate the pharmacokinetics of a single dose of 1500 mg (2 x 750 mg), a single dose of 2250 mg (3 x 750 mg), and a single dose of 3000 mg (4 x 750 mg) gepotidacin tablet formulation (RC or HSWG tablet) selected from Part 1a or placebo under fed conditions.

#### Dosing

## Part 1a - Relative Bioavailability:

- Treatment A: Gepotidacin 1500 mg (3 × 500 mg) reference capsules
- Treatment B: Gepotidacin 1500 mg (2 × 750 mg) RC tablets
- Treatment C: Gepotidacin 1500 mg (2 × 750 mg) HSWG tablets

## Part 1b (Optional) – Food Effect:

- Treatment D: Gepotidacin 1500 mg (2 × 750 mg) RC or HSWG tablets selected from Part 1a – fasted
- Treatment E: Gepotidacin 1500 mg (2 × 750 mg) RC or HSWG tablets selected from Part 1a – fed

## Part 2: Pharmacokinetics in Japanese Subjects

- Treatment B or C: Gepotidacin 1500 mg (2 × 750 mg) RC (Treatment B) or HSWG (Treatment C) tablets selected from Part 1a – fasted
- Treatment F: Gepotidacin 3000 mg (4 × 750 mg) RC or HSWG tablets selected from Part 1a – fasted

## Part 3: Pharmacokinetics in Japanese Subjects – Fed State

- Treatment E: Gepotidacin 1500 mg (2 × 750 mg) RC or HSWG tablets selected from Part 1a – fed
- Treatment G: Gepotidacin 2250 mg (3 × 750 mg) RC or HSWG tablets selected from Part 1a – fed
- Treatment H: Gepotidacin 3000 mg (4 × 750 mg) RC or HSWG tablets selected from Part 1a – fed
- Treatment I: Placebo tablets fed

# Treatment Assignment

- Part 1a Relative Bioavailability: On Day 1 (Period 1), subjects will be randomly assigned to a treatment sequence (ABC, CAB, or BCA) to receive a single dose of gepotidacin 1500 mg (2 × 750 mg) RC tablet,1500 mg (2 × 750 mg) HSWG tablet, or 1500 mg (3 × 500 mg) reference capsule under fasted conditions in each period.
- Part 1b (Optional) Food Effect: On Day 1 (Period 1), subjects will be randomly assigned to a treatment sequence (DE or ED) and receive a single 1500 mg (2 × 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a under fasted and fed conditions.
- Part 2 Pharmacokinetics in Japanese Subjects: On Day 1 of Period 1,

| Overview of | Study Design and Key Features |
|---|---|
| | subjects will receive a single 1500 mg (2 × 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a under fasted conditions. On Day 1 of Period 2, subjects will receive a single 3000-mg (4 × 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a under fasted conditions. |
| | Part 3 – Pharmacokinetics in Japanese Subjects – Fed State: On Day 1 (Period 1), subjects will be stratified by gender, randomized to active or placebo in a 5:1 ratio to receive gepotidacin tablet (RC or HSWG) selected from Part 1a in an ascending manner (Treatments E, G, and H) on Day 1 of Period 1, 2, and 3, respectively, or placebo (Treatment I). For each period, a sentinel group of up to four subjects will be dosed with study drug and evaluated for safety and tolerability prior to dosing remaining subjects. |
| Interim<br>Analysis | <ul> <li>No formal interim analyses are planned for this study. However, all preliminary safety, tolerability, and available PK data will be reviewed by the study team after completing Part 1a of the study to select the formulation for Part 1b, Part 2, and Part 3, and also to determine if the effect of food on the selected formulation needs to be studied (Part 1b). The team will review unblinded data from Part 1a of this open-label study to select the appropriate formulation.</li> </ul> |

## 2.4. Statistical Hypotheses

A formal hypothesis will not be tested; however, an estimation approach will be taken to characterize the bioavailability of the gepotidacin RC and HSWG tablet formulations relative to the reference gepotidacin capsule formulation in healthy subjects (Part 1a), estimate the effect of food on the tablet formulation selected in Part 1a (Part 1b), and to evaluate the pharmacokinetics of the tablet formulation selected in Part 1a in Japanese subjects (Parts 2 and 3).

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No formal interim analyses are planned for this study. However, all preliminary safety, tolerability, and available PK data will be reviewed by the study team after completing Part 1a of the study to select the formulation for Part 1b, Part 2, and Part 3, and also to determine if the effect of food on the selected formulation needs to be studied (Part 1b). The team will review unblinded data from Part 1a of this open-label study to select the appropriate formulation.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

1. All subjects have completed the study as defined in the protocol.

2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Safety Population | Will consist of all subjects who receive at least<br>1 dose of study drug and have at least 1 post<br>dose safety assessment. | <ul><li>Study Population</li><li>Safety</li></ul> |
| | This population will be based on the treatment which the subject actually received. | |
| PK Population | Will consist of all subjects who received at least 1 dose of gepotidacin and have evaluable PK data for gepotidacin. | PK Concentration |
| PK Parameter<br>Population | Will consist of all subjects in the PK Population, for whom valid and evaluable PK parameters were derived. This population will be used in the assessment and characterization of PK parameters. | PK Parameters |

#### NOTES:

Please refer to Appendix 11 which details the population to be used for each display being generated.

## 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States and Phases |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Division of Microbiology and Infectious Disease Adult Toxicity Tables for Adverse Event Assessment |
| 10.8 | Appendix 8: Multiple Comparisons and Multiplicity |
| 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| 10.10 | Appendix 10: Abbreviations & Trade Marks |
| 10.11 | Appendix 11: List of Data Displays |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Display's Generated | | |
|---|---|---|---|
| | Figure | Table | Listing |
| Enrollment | | | |
| Number of Subjects Enrolled by Country and Site ID | | Υ | |
| Randomisation | | | |
| Randomisation | | | Υ |
| Subject Disposition | | | |
| Subject Disposition | | Υ | |
| Reasons for Screening Failures | | Υ | Υ |
| Reasons for Withdrawals | | | Υ |
| Important Protocol Deviations | | Υ | Υ |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Demography | | | |
| Demographics Characteristics | | Y | Y |
| Study Populations | | | Υ [1] |
| Medical Condition & Concomitant Medications | | | |
| Medical Conditions (Current/Past) | | | Y |
| Concomitant Medication | | | Y |

#### NOTES:

- Y = Yes display generated.
- 1. Listing of subjects excluded from any population will be generated only.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Pharmacokinetic Analyses

## 7.1.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK Population for plasma PK concentrations, and PK Parameter Population for plasma/urine PK parameters, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Display Type | | Untransformed | | | | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis Summary | | mary | Individual | | Stats Analysis | | Summary | | Individual | | | |
| | Т | F | L | Τ | F | F | L | Т | F | L | Т | F | F | L |
| Plasma PK | | | | V | <b>Y</b> [1] | <b>Y</b> [1] | ٧ | | | | | <b>Y</b> [1] | <b>Y</b> [1] | |
| Concentrations | | | | I | [2] | 11.1 | I | | | | | [2] | 11.1 | |
| Urine PK | | | | V | <b>Y</b> [1] | <b>Y</b> [1] | ٧ | | | | | <b>Y</b> [1] | <b>Y</b> [1] | |
| Concentrations | | | | ľ | [2] | 1 L L L L L L L L L L L L L L L L L L L | ľ | | | | | [2] | 1,11 | |
| Plasma PK | <b>&gt;</b> | <b>&gt;</b> | | V | | | V | <b>&gt;</b> | | | V | | \<br>\ | |
| Parameters | ı | ı | | I | | | I | ı | | | I | | ı | |
| Urine PK Parameters[3] | | | | Υ | | | Υ | | | | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Linear and Semi-Log plots will be created on the same display.
- [2] Separate mean and median plots will be generated.
- [3] Parts 1a, 2 and 3 only.

## 7.1.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 3 Reporting Process & Standards).

#### 7.1.3. Pharmacokinetic Parameters

## 7.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 3 Reporting Process & Standards).
- The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.

- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 4 will be determined from the plasma concentration-time data, as data permits.
- Pharmacokinetic parameters described in Table 5 will be determined from the urine concentration data, as data permits.

 Table 4
 Derived Plasma Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve (AUC) from time 0 (predose) to time of the last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, calculated as: |
| | $AUC(0-\infty) = AUC(0-t) + C(t) / \lambda z$ |
| | where C(t) is the last observed quantifiable concentration. |
| %AUCex | The percentage of AUC (0-∞) obtained by extrapolation (%AUCex) will be calculated as: |
| | [AUC(0-∞) – AUC(0-t)] / AUC(0-∞) x 100 |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to first occurrence of Cmax |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| t½ | Terminal phase half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| Frel | Relative bioavailability of drug, calculated as: |
| | Frel = $[AUC(0-\infty)_{tablet}]/[AUC(0-\infty)_{capsule}]$ (Part 1a only) |
| λz | Terminal-phase rate constant |
| DNAUC(0-t) | Dose normalized area under the concentration-time curve from time 0 (predose) to time of the last quantifiable concentration (Part 2 and Part 3 for use in the pooled analysis with Part 2), to be calculated as |
| | DNAUC(0-t) = AUC(0-t) / Dose |
| DNAUC(0-∞) | Dose normalized area under the concentration-time curve from time 0 (predose) extrapolated to infinite time (Part 2 and Part 3 for use in the pooled analysis with Part 2), calculated as: |
| | $DNAUC(0-\infty) = AUC(0-\infty) / Dose$ |
| DNCmax | Dose normalized maximum observed concentration (Part 2 and Part 3 for use in the pooled analysis with Part 2), to be calculated as |

| Parameter | Parameter Description | |
|-----------|-----------------------|----------------------|
| | | DNCmax = Cmax / Dose |

## NOTES:

• Additional parameters may be included as required.

## Table 5 Derived Urine Pharmacokinetic Parameters (Parts 1a, 2, and 3 only)

| Parameter | Parameter Description |
|---|---|
| Ae total | Total unchanged drug (total amount of drug excreted in urine), calculated by adding all the fractions of drug collected over all the allotted time intervals |
| Ae(t1-t2) | Amount of drug excreted in urine in a time intervals for predose, 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours. |
| AUC(0-12) | Area under the urine concentration-time curve over time 0 (predose) to 12 hours after dosing. The AUC will be calculated by the linear trapezoidal rule based on the urine concentration data from each collection interval versus the corresponding urine collection interval. |
| AUC(0-24) | Area under the urine concentration-time curve over time 0 (predose) to 24 hours after dosing. The AUC will be calculated by the linear trapezoidal rule based on the urine concentration data from each collection interval versus the corresponding urine collection interval. |
| AUC(0-48) | Area under the urine concentration-time curve over time 0 (predose) to 48 hours after dosing. The AUC will be calculated by the linear trapezoidal rule based on the urine concentration data from each collection interval versus the corresponding urine collection interval. |
| fe% | Percentage of the given dose of drug excreted in urine, calculated as: |
| | fe% = (Ae total/Dose) × 100 |
| CLr | Renal clearance of drug, calculated as: |
| | CLr = Ae total/AUC(0-t) |

## NOTES:

• Additional parameters may be included as required.

# 7.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

The following PK statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

| Pharmacokinetic Statistical Analyses | |
|---|---|
| Endpoint(s) | |
| <ul> <li>Plasma primary PK endpoints include AUC(0-∞), AUC(0-t) and Cmax of gepotidacin,<br/>data permit</li> </ul> | as |
| Model Specification | |
| • The log-transformed AUC(0-∞), AUC(0-t), and Cmax values for gepotidacin will be analyzed | ed |

## **Pharmacokinetic Statistical Analyses**

separately using a mixed effects model as appropriate to the study design, fitting fixed effect terms for sequence, period, and regimen, and treating subject within sequence as a random effect. Point estimates and 90% confidence intervals (CIs) for the differences of interest (RC tablets and HSWG tablets versus capsules) will be constructed using the residual variance

- In the optional food effects study in Part 1b, the log-transformed AUC(0-∞), AUC(0-t), and Cmax values for gepotidacin will be analyzed separately using a mixed effects model as appropriate to the study design, fitting fixed effect terms for sequence, period, and regimen, and treating subject within sequence as a random effect. Point estimates and 90% CIs for the differences of interest (tablet formulation under fasted and fed conditions) will be constructed using the residual variance. The ratio of geometric mean and 90% CIs of ratio will be obtained by exponentiation of the point estimates and 90% CIs for the difference on the natural logarithmic scale.
- For the bioavailability assessment, Tmax will be analyzed nonparametrically using the Wilcoxon signed-rank test to compute the point estimate and 90% CI for the median difference for each comparison of interest.
- In Part 2, dose proportionality will be evaluated for the dose-normalized (DN) PK parameters for gepotidacin: DNAUC(0-∞), DNAUC(0-t), and DNCmax. An analysis of variance (ANOVA) model with log transformed DN PK parameters [DNAUC(0-∞), DNAUC(0-t), and DNCmax] as dependent variable, dose group as a fixed effect and subject as a random effect will be used to estimate the DN geometric means of each dose, and the ratio of geometric means between two doses (3000 mg vs 1500 mg) with 90% CI for Part 2 subjects alone. Additionally, subjects in Part 2 (fasted) and Part 3 (fed) will be pooled together in an exploratory analysis to assess the dose proportionality between 3000 mg and 1500 mg. There would be evidence of dose proportionality if the 90% CI for the ratio of DN geometric means lies within the limits (0.80, 1.25).
- For Parts 2 and 3, PK parameters will be summarized based on pooled data (for the doses (1500 mg and 3000 mg).
- Additionally, for Part 3, dose proportionality in the Japanese fed cohort portion of the study will be evaluated by using the power model:

$$y = \alpha \times (dose)^{\beta}$$

where y denotes the PK parameter being analyzed [AUC(0- $\infty$ ), AUC(0-t), and Cmax]. Dose proportionality implies that  $\beta$  = 1 and will be assessed by estimating  $\beta$  along with its 90% confidence interval. The exponent,  $\beta$ , in the power model will be estimated by regressing the natural log-transformed PK parameter on natural log-transformed dose.

$$Ln(y)=In(\alpha) + \beta * In(dose)$$

The power model will be fitted by restricted maximum likelihood (REML) using SAS Proc Mixed with subject as a random effect, or a fixed effect power model will be fitted. The mean slope will be estimated from the power model and the corresponding 90% confidence interval calculated. Point estimates and confidence intervals for the slope will be reported to 4 decimal places with no rounding.

## **Pharmacokinetic Statistical Analyses**

PK parameters for all subjects will be evaluated using the Grubbs' test [Grubbs, 1950] on the
natural log-transformed PK parameters by treatment. For study parts where subjects have
been identified as outliers, additional analyses will be performed with outliers excluded.

## **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Statistical analysis by analysis of variance (ANOVA) will be presented in tabular format with geometric mean ratios between RC tablets and HSWG tablets versus capsules, and 90% CIs for the ratios of AUC(0-∞) and Cmax for gepotidacin.
 Example SAS Code:

PROC MIXED:

CLASS USUBJID TRTA TRTSEQP APERIOD:

MODEL LOGPKPARM =TRTA TRTSEQP APERIOD /DDFM=KR;

RANDOM USUBJID(TRTSEQP);

LSMEANS TRTA;

ESTIMATE 'B VS A' TRTA -1 1 0/CL ALPHA=0.1;

ESTIMATE 'C VS A' TRTA -1 0 1/CL ALPHA=0.1;RUN;

 Statistical analysis by ANOVA for the optional food effect (Part 1b) will be presented in tabular format with geometric mean ratios between tablet formulation under fasted and fed conditions, and 90% CIs for the ratios of AUC(0-∞) and Cmax for gepotidacin.
 Example SAS Code:

PROC MIXED:

CLASS USUBJID TRTA TRTSEQP APERIOD;

MODEL LOGPKPARM =TRTA TRTSEQP APERIOD /DDFM=KR;

RANDOM USUBJID(TRTSEQP);

LSMEANS TRTA;

ESTIMATE 'E VS D' TRTA -1 1/CL ALPHA=0.1; RUN;

 Statistical analysis of Tmax will be analyzed nonparametrically using the Wilcoxon signed-rank test.

Example SAS Code:

PROC UNIVARIATE DATA=PK WILCOXON;

VAR DIFF: /\*DIFFERENCE OF AVAL FOR TREATMENT A-B \*/

CLASS TRTA;

ODS OUTPUT =PVAL;

RUN;

• Statistical analysis by ANOVA for Part 2 and Part 3 will be presented in tabular format with geometric mean ratios between 3000-mg and 1500-mg (Part 2 alone and Parts 2 and 3 pooled), and 90% CIs for the ratios of DNAUC(0-t), DNAUC(0-∞) and DNCmax for gepotidacin.

Example SAS Code:

## Pharmacokinetic Statistical Analyses

ODS OUTPUT LSMEANS=LSM DIFFS=PAIR;

PROC MIXED DATA=PK3:

CLASS USUBJID DOSE:

MODEL LOGPP=DOSE/SOLUTION ALPHA=0.1 CL DDFM=KR;

RANDOM SUBJECT;

LSMEANS DOSE/PDIFF(CONTROL='1500 mg') ALPHA=0.1 CL;

RUN:

 Statistical analysis by REML for the Japanese food effect (Part 3) will be presented in tabular format to present the exponent β and 90% CI for the AUC(0-∞), AUC(0-t), and Cmax for gepotidacin in fed Japanese subjects.

Example SAS Code:

PROC MIXED;

CLASS SUBJECT:

MODEL LOGPKPARM =LOGDOSE /CL ALPHAS-0.1 SOLUTION;

RUN;

## 7.1.4. Interim Analysis

## 7.1.4.1. Overview of Planned Analyses

Interim analysis is planned for Part 1a. Available PK data will be reviewed by the study team after completing Part 1a of the study to select the formulation for Part 1b, Part 2, and Part 3, and also to determine if the effect of food on the selected formulation needs to be studied (Part 1b).

Table 7 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Plasma concentrations of gepotidacin will be subjected to PK analyses using noncompartmental methods. Based on the individual concentration time data the following parameters will be estimated:

Table 6 Derived Plasma Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time 0 (predose) to time of the last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, calculated as: |
| | $AUC(0-\infty) = AUC(0-t) + C(t) / \lambda z$ |
| | where C(t) is the last observed quantifiable concentration. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to first occurrence of Cmax |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| t½ | Terminal phase half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| Frel | Relative bioavailability of drug, calculated as: |
| | Frel = $[AUC(0-\infty)]$ tablet]/[ $AUC(0-\infty)$ capsule] (Part 1a only) |

## NOTES:

Additional parameters may be included as required.

The log-transformed AUC( $0-\infty$ ), AUC(0-t), and Cmax values for gepotidacin will be analyzed separately using a mixed effects model as appropriate to the study design, fitting fixed effect terms for sequence, period, and regimen, and treating subject within sequence as a random effect (Section 7.1.3.2).

For the bioavailability assessment, Tmax will be analyzed nonparametrically using the Wilcoxon signed-rank test to compute the point estimate and 90% CI for the median difference for each comparison of interest (Section 7.1.3.2).

Table 7 provides an overview of the planned interim analyses.

Table 7 Overview of Planned Interim Analyses

| Display Type | | Untransformed | | | | | | | | Log-Transformed | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Anal | lysis | Sumi | Summary Individual | | | Stat | s Anal | ysis | Summary | | Individual | |
| | Т | F | L | T | F | F | Ш | T | F | L | T | F | F | Ш |
| Plasma PK | | | | V | <b>Y</b> [1] | <b>Y</b> [1] | ٧ | | | | V | <b>Y</b> [1] | <b>Y</b> [1] | |
| Concentrations | | | | I | [2] | 11.1 | ı | | | | I | [2] | 11.1 | |
| Urine PK | | | | V | <b>Y</b> [1] | <b>Y</b> [1] | <b>&gt;</b> | | | | V | <b>Y</b> [1] | <b>Y</b> [1] | |
| Concentrations | | | | I | [2] | 11.1 | ı | | | | I | [2] | 11.1 | |
| Plasma PK | V | | | V | | | V | <b>V</b> | | | V | | | |
| Parameters | I | | | I | | | I | Ī | | | T | | | |
| Urine PK Parameters | | | | Υ | | | Υ | | | | Υ | | | |

## NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Linear and Semi-Log plots will be created on the same display.
- [2] Separate mean and median plots will be generated.

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Safety Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 8 provides an overview of the planned safety analyses with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 8 Overview of Planned Safety Analyses

| Display Type | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | nmary | Indiv | /idual | Sum | mary | Indiv | /idual |
| | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Extent of Exposure | | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| All AEs | Υ | | | Y | | | | |
| All Drug-Related AEs | Υ | | | Y | | | | |
| Serious AEs | Υ | | | Υ | | | | |
| Withdrawal AEs | | | | Υ | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | | | | Υ | Υ | | | |
| Hematology | | | | Υ | Y | | | |
| Urinalysis (Dipstick) | Υ | | | Υ | | | | |
| ECGs | | | | | | | | |
| ECG Findings | Υ | | | Υ | | | | |
| ECG Values | | | | Υ | Y | | | Υ |
| Vital Signs | | | | | | | | |
| Vital Signs | | | | Υ | Υ | | | |
| Liver | | | | | | | | |
| Liver Events [1] | | | | Υ | | | | |
| Cardiovascular | | | | | | | | |
| Cardiovascular [1] | | | | Y | | | | |
| Clostridium Difficile | | | | | | | | |
| Clostridium difficile | | | | Y | | | | |
| Testing [1] | | | | | | | | |
| Rash Events | | | | | | | | |
| Rash Events [1] | | | | Y | | | | |
| NOTES · | | | | 1 | 1 | | | <u> </u> |

#### NOTES:

- 1. Conditional displays, they will only be produced when an event has occurred.
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual subject observed raw data.

## 9. REFERENCES

GlaxoSmithKline Document Numbers 2016N281831\_02 (Original – 12-JUL-2016): A Phase I; Multi-Center; Open-Label (Parts 1 and 2); Randomized, Double-Blind, Placebo-Controlled (Part 3); Single-Dose, 3-Part Study to Evaluate the Relative Bioavailability of Three Formulations in Healthy Subjects, Food Effect on Tablet Formulation in Healthy Subjects, and Pharmacokinetics of Gepotidacin (GSK2140944) in Japanese Subjects in Fasted and Fed States (05-SEP-2017)

Grubbs FE. Sample Criteria for Testing Outlying Observations, Annals of Math. Statistics 1950, 21: 27-58.

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5: | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States & Phases |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7: Division of Microbiology and Infectious Disease Adult Toxicity Tables |
| 0 " 10 0 | for Adverse Event Assessment |
| Section 10.8 | Appendix 8: Multiple Comparisons and Multiplicity |
| Section 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |

# 10.1. Appendix 1: Time & Events

## 10.1.1. Protocol Defined Time & Events

Time and Events Table: Parts 1a. 1b. 2a. 2b. and 3

| Time and Events Table: Parts 1a, 1 | b, 2a, 2b, and | 13 | • | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | Pa | Part 1b<br>rt 2 - Ph | - Food<br>narmaco | Effect:<br>okinetio | Periods | s 1 and<br>ods 1 a | | | | | | Follow-<br>up (5 to |
| Procedure | (up to 30 days prior | Day<br>-1ª | | | | | | | Day 1 | | | | | | Da | y 2 | Day<br>3 | 7 days<br>post-last |
| | to Day 1) | | Pre-dose | 0h | 0.5 h | 1 h | 1.5 h | 2 h | 2.5 h | 3 h | 4 h | Ч9 | 8 h | 12 h | 24 h | 36 h | 48 h | dose) |
| Admission to Unit | | Х | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Demographics including BMI | X | | | | | | | | | | | | | | | | | |
| Full physical examination including height and weight <sup>b</sup> | x | | | | | | | | | | | | | | | | | |
| Brief physical examination <sup>b</sup> | | Х | | | | | | | | | | | | | | | | Х |
| Medical/medication/drug/alcohol history | x | | | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>c</sup> | Х | Х | Х | | | | | Х | | | | | | | Х | | Х | Х |
| Vital signs <sup>d</sup> | Х | Х | Χ | | | | | Χ | | | | | | | Χ | | Х | Х |
| Drug/alcohol/cotinine screen | X | Х | | | | | | | | | | | | | | | | |
| Serum pregnancy, FSH, and estradiol (women) | х | Х | | | | | | | | | | | | | | | | х |
| HIV antibody, HBsAg, and hepatitis C antibody screen | х | | | | | | | | | | | | | | | | | |
| Safety laboratory tests <sup>e</sup> | Х | Х | | | | | | | | | | | | | | | Х | Х |
| Study drug administration <sup>f</sup> | | | | Х | | | | | | | | | | | | | | |
| Pharmacokinetic sampling | | | Х | | Х | Χ | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | |
| Urine collection for pharmacokinetics (Parts 1a, 2, and 3 only) <sup>g</sup> | | | Х | | | | | | Х | | Х | Х | Х | Х | Х | Х | Х | |

Time and Events Table: Parts 1a, 1b, 2a, and 2b, cont.

| Time and Events | | , -, -, - | , | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | Part 1a - Relative Bioavailability: Periods 1, 2, and 3 Part 1b - Food Effect: Periods 1 and 2 Part 2 - Pharmacokinetics: Periods 1 and 2 | | | | | | | | | | | | | | |
| Procedure | days prior to | | | Day 1 Day 2 3 | | | | | | | | | | | | Follow-up (5 to 7 days post-<br>last dose) | | |
| Day 1) | рау 1) | Day 1) | Pre-dose | 0h | 0.5 h | 1 h | 1.5 h | 2 h | 2.5 h | 3 h | 4 h | 6 h | 8 h | 12 h | 24 h | 36 h | 48 h | |
| Pharmacogenetic sample <sup>h</sup> | | | | | | + | -==== | | | ===== | | | ===== | | => | | | |
| AE/SAE Review | Х | | | <b>←===</b> | ===== | | ===== | | ===== | | ===== | ===== | | ===== | $\rightarrow$ | | | X |
| Concomitant<br>medication<br>review | | Х | | ←=====→ | | | | | | | | Х | | | | | | |
| Discharge <sup>i</sup> | | | | | | | | | | | | | | | | | Х | |
| Outpatient visit | Х | | | | | | | | | | | | | | | | | X |

AE = adverse event, BMI = body mass index, ECG = electrocardiogram, FSH = follicle-stimulating hormone, HBsAg = hepatitis B surface antigen, HIV = human immunodeficiency virus, SAE = serious adverse event

The Day -1 visit occurs in Period 1 only. Periods 2 (all parts) and 3 (Parts 1a and 3 only) begin on Day 1.

A complete physical examination will include at a minimum, assessment of the cardiovascular, respiratory, GI, and neurological systems. Height and weight will also be measured and recorded. A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen)

Triplicate 12-lead ECGs will be measured in semi-supine position after 5 minutes rest and obtained at least 5 minutes apart on Day -1. Single 12-lead ECGs will be measured in semi-

supine position after 5 minutes rest at all other time points during the study.

Single vital signs will be measured in semi-supine position after 5 minutes rest and will include systolic and diastolic blood pressure, and heart rate. Body temperature and

respiratory rate will be collected at Screening only.

Safety laboratory tests include serum chemistry, hematology, and urinalysis.

Subjects will fast from food and drink (except water) for at least 10 hours before study drug administration on Day 1 of each period. For the fed group of the food effect evaluation in Part 1b, study drug will be administered within 30 minutes after the completion of a moderate fat meal. For Part 3, study drug will be administered within 30 minutes after completion of a standard Japanese meal.

Urine collection intervals (Parts 1a, 2 and 3 only) for subjects include 0 (pre-dose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours.

For subjects who consent only: collect 1 pharmacogenetic sample after the start of dosing (preferably Day 1). Informed consent for optional pharmacogenetic research must be obtained before collecting a sample.

For Parts 1a and 3, subjects will be discharged from the clinic research unit on Day 3 of Period 3. For Parts 1b and 2, subjects will be discharged on Day 3 of Period 2.

# 10.2. Appendix 2: Treatment States and Phases

## 10.2.1. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment for the respective treatment period.

## 10.2.1.1. Treatment States for Safety Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date/Time < Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time ≤ Date/Time ≤ Study Treatment Stop Date/Time + 2 Days |
| Post-Treatment | Date/Time > Study Treatment Stop Date/Time +2 Days |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

## 10.2.1.2. Treatment States for AE Data

| Treatment<br>State | Definition |
|---|---|
| Pre-Treatment | AE Start Date/Time < Study Treatment Start Date/Time |
| On-Treatment | If AE onset date/time is on or after treatment start date/time & on or before the treatment stop date/time with 2 days lag time |
| On-Treatment | Study Treatment Start Date/Time ≤ AE Start Date/Time ≤ Study Treatment Stop Date/Time + 2 Days |
| Post Treatment | If AE onset date/time is after the treatment stop date/time with 2 days lag time |
| Post-Treatment | AE Start Date/Time > Study Treatment Stop Date/Time + 2 days |
| Onset Time | If Treatment Start Date/Time > AE Onset Date/Time = AE Onset Date - Treatment Start Date |
| Since First Dose | If Treatment Start Date/Time ≤ AE Onset Date/Time = AE Onset Date - Treatment Start |
| (Days) | Date +1 |
| | Missing otherwise |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

## 10.3.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | | |
|---|---|---|---|---|
| Study | | Treatment Group | Data Displays for Report | ing |
| Part | Code | Description | Description | Order [1] |
| 1a | А | Gepotidacin 1500 mg (3 × 500 mg) reference capsules | Reference | 1 |
| 1a, 2 <sup>[3]</sup> | В | Gepotidacin 1500 mg (2 × 750 mg)<br>RC tablets | RC 1500 mg | 2 |
| 1a, 2 <sup>[3]</sup> | С | Gepotidacin 1500 mg (2 × 750 mg)<br>HSWG tablets | HSWG 1500 mg | 3 |
| 1b | D | Gepotidacin 1500 mg (2 × 750 mg) | RC 1500 mg Fasted or | 4 |
| | | RC or HSWG tablets selected from Part 1a – fasted | HSWG 1500 mg Fasted <sup>[2]</sup> | |
| 1b, 3 | Е | Gepotidacin 1500 mg (2 × 750 mg) | RC 1500 mg Fed or | 5 |
| | | RC or HSWG tablets selected from Part 1a – fed | HSWG 1500 mg Fed <sup>[2]</sup> | |
| 2 | F | Gepotidacin 3000 mg (4 × 750 mg) | RC 3000 mg or | 6 |
| | | RC or HSWG tablets selected from Part 1a | HSWG 3000 mg <sup>[2]</sup> | |
| 3 | G | Gepotidacin 2250 mg (3 × 750 mg) | RC 2250 mg Fed or | 7 |
| | | RC or HSWG tablets selected from Part 1a – fed | HSWG 2250 mg Fed <sup>[2]</sup> | |
| 3 | Н | Gepotidacin 3000 mg (4 × 750 mg) | RC 3000 mg Fed or | 8 |
| | | RC or HSWG tablets selected from Part 1a – fed | HSWG 3000 mg Fed <sup>[2]</sup> | |
| 3 | ı | Placebo | Placebo | 9 |

#### NOTES:

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. The use of "RC" vs "HSWG" will be determined after study part 1a.
- 3. In part 2, one of Treatment B or Treatment C (determined after study part 1a) will be administered in period 1.

## 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

For all endpoints (expect as noted in the table) the baseline value will be the latest predose assessment and are applicable to each period.

Table 9 Baseline Definitions

| Parameter | Study Assess | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Data Display | |
| Safety | | | | |
| Hematology | X | Χ | | Day -1 |
| Clinical Chemistry | X | Χ | | Day -1 |
| 12 Lead ECG | Х | Х | Х | Day 1 (Pre-dose) |
| Vital Signs | X | Χ | X | Day 1 (Pre-dose) |

#### NOTES:

 Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

## 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 10.3.3. Reporting Process & Standards

#### Reporting Process

#### Software

The currently supported versions of SAS and WinNonlin software will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & ADaM IG Version 1.0].
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

## **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables

## **Reporting Standards**

7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

## **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### Unscheduled Visits

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| 7 th dhoshedded visits will be moldded in nothings. | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | NQs at the beginning of a subject profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood. |
| | <ul> <li>For NQs at the end of the subject profile (i.e. after the last incidence<br/>of a measurable concentration);</li> </ul> |
| | <ul> <li>for individual plots and pharmacokinetic analyses these are<br/>dropped (set to missing) as they do not provide any useful</li> </ul> |

| Reporting Standards | Reporting Standards |
|---|---|
| | information (and can erroneously indicate that absolutely no drug is present) |
| | <ul> <li>for summary statistics these are set to 0 (to avoid skewing of the<br/>summary statistics)</li> </ul> |
| | <ul> <li>Individual NQs which fall between two measurable concentrations<br/>are set to missing (individual values of this nature are assumed to be<br/>an anomaly)</li> </ul> |
| | <ul> <li>If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual subject plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).</li> </ul> |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive Summary<br>Statistics.<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between subject coefficient of variation (CVb (%)) will be reported. |
| | CVb (%) = $\sqrt{(\exp(SD^2) - 1) * 100}$ [NOTE: SD = SD of log transformed data] |
| Parameters Not Being<br>Log Transformed | Tmax, first point, last point and number of points used in the determination of $\lambda z$ . |
| Parameters Not Being<br>Summarised | Additionally include tmax, first point, last point and number of points used in the determination of $\lambda z$ . |
| Listings | Include the first point, last point and number of points used in the determination of $\lambda z$ . |
| <b>Graphical Displays</b> | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 10.4. Appendix 4: Derived and Transformed Data

## 10.4.1. **General**

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## Study Day

- Calculated as the number of days from randomisation date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

## 10.4.2. Study Population

## **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date is imputed as:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

## 10.4.3. Safety

#### **ECG Parameters**

#### RR Interval

- If ECG values are machine read and either RR interval (msec) is not provided directly, then these can be derived as:
  - [1] If QTcB is machine read & RR is not provided, then:

## **ECG Parameters**

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and RR is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^3 \right] * 1000$$

- If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.
- Important Note: Machine read values of RR should not be replaced with derived values.

#### Corrected QT Intervals

- When not entered directly in the eCRF, corrected QT intervals using Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}} \qquad \qquad QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

Important Note: Machine read values of QTcB and QTcF should not be replaced with rederived values. If neither machine read QTcB or QTcF are available but QT and RR are
collected, then a QTcB and QTcF can be derived however this should be discussed and
agreed with the study team and the TLFs must have an appropriate footnote denoting those
parameters are derived.

#### **Adverse Events**

## **AE's of Special Interest**

- Liver events
- Cardiovsacular events
- Potential systemic allergic reactions
- Gl events
- Acetylcholinesterase (AChE) Inhibition

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

## 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument : |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | <ul> <li><u>Missing Start Day:</u> First of the month will be used unless this is before the<br/>start date of investigational product; in this case the study treatment start<br/>date will be used (and hence the event is considered On-treatment as per<br/>Appendix 2: Treatment States and Phases).</li> </ul> |
| | <ul> <li><u>Missing Stop Day</u>: Last day of the month will be used, unless this is after the<br/>stop date of study treatment; in this case the study treatment stop date will<br/>be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation |

| Element | Reporting Detail |
|---|---|
| | applied. Consequently, time to onset and duration of such events will be missing. |
| | Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied. |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month.</li> </ul> |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event<br/>could possibly have occurred during treatment from the partial information,<br/>then the Week 1 Day 1 date will be assumed to be the start date.</li> </ul> |
| | <ul> <li>The AE will then be considered to start on-treatment (worst case).</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. ECG

| ECG Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450[1] | |
| Absolute OTe Intervel[3] | maaa | > 450[2] | ≤ 479 <sup>[2]</sup> |
| Absolute QTc Interval <sup>[3]</sup> | msec | ≥ 480 <sup>[2]</sup> | ≤ 499 <sup>[2]</sup> |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110[1] | > 220[1] |
| Absolute QRS Interval | msec | < 75[1] | > 110[1] |
| Change from Baseline | | | |
| | msec | ≤ 30[2] | |
| Increase from Baseline QTc[3] | msec | > 30[2] | ≤ 59 <sup>[2]</sup> |
| | msec | ≥ 60[1] | |

#### NOTES:

- 1. Represent standard ECG values of PCI for HV studies.
- Represent further subdivisions of ECG values for analysis.
- 3. Qualifying QTc events, regardless whether QTcB or QTcF, will be captured.

# 10.6.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7: Division of Microbiology and Infectious Disease Adult Toxicity Tables for Adverse Event Assessment

# 10.7.1. Laboratory Values

Parameter values are converted to use SI units.

#### HEMATOLOGY

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hemoglobin | 95 to 105 G/L | 80 to 94 G/L | 65 to 79 G/L | <65 G/L |
| Absolute neutrophil count | 1.0 to 1.5 10^9/L | 0.75 to 0.999 10^9/L | 0.5 to 0.749 10^9/L | <0.5 10^9/L |
| Platelets | 75 to 99.999 10^9/L | 50 to 74.999 10^9/L | 20 to 49.999 10^9/L | <20 10^9/L |
| White Blood Cells | 11 to 13 10^9/L | 13 to 15 10^9/L | 15 to 30 10^9/L | >30 or <1 10^9/L |
| % Polymorphonuclear leukocytes + band cells | >80% | 90 to 95% | >95% | N/A |
| Abnormal Fibrinogen | Low: 1 to 2 G/L<br>High: 4 to 6 G/L | Low: <1 G/L<br>High: >6 G/L | Low: <0.5 G/L<br>High: N/A | Fibrinogen associated with gross bleeding or with disseminated coagulation |
| Fibrin Split Product | 0.020 to 0.040 G/L | 0.041 to 0.050 G/L | 0.051 to 0.060 G/L | >0.060 G/L |
| Prothrombin Time | 1.01 to 1.25 × ULN | 1.26 to 1.5 × ULN | 1.51 to 3.0 × ULN | >3 × ULN |
| Activated Partial Thromboplastin | 1.01 to 1.66 × ULN | 1.67 to 2.33 × ULN | 2.34 to 3 × ULN | >3 × ULN |
| Methemoglobin | 5.0 to 9.9% | 10.0 to 14.9% | 15.0 to 19.9% | >20% |
| N/A = not applicable; ULN = upper limit of | normal. | | | |

#### CHEMISTRIES

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hyponatremia | 130 to 135 MMOL/L | 123 to 129 MMOL/L | 116 to 122 MMOL/L | <116 MMOL/L or abnormal sodium with |
| Туропанстна | 100 to 100 MINIOL/E | 123 to 123 WINDE/E | 110 to 122 WINIOL/E | mental status changes or seizures |
| Hypernatremia 1 | 146 to 150 MMOL/L | 151 to 157 MMOL/L | 158 to 165 MMOL/L | >165 MMOL/L or abnormal sodium with |
| | | | | mental status changes or seizures |
| Hypokalemia | 3.0 to 3.4 MMOL/L | 2.5 to 2.9 MMOL/L | 2.0 to 2.4 MMOL/L or intensive replacement therapy of hospitalization required | <2.0 MMOL/L or abnormal potassium with paresis, ileus, or life-threatening arrhythmia |

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hyperkalemia | 5.6 to 6.0 MMOL/L | 6.1 to 6.5 MMOL/L | 6.6 to 7.0 MMOL/L | >7.0 MMOL/L or abnormal potassium with life-threatening arrhythmia |
| Hypoglycemia | 3.0 to 3.55 MMOL/L | 2.22 to 2.99 MMOL/L | 1.67 to 2.21 MMOL/L | <1.67 MMOL/L or abnormal glucose with mental status changes or coma |
| Hyperglycemia<br>(nonfasting and no prior<br>diabetes) | 6.44 to 8.88 MMOL/L | 8.89 to 13.88 MMOL/L | 13.89 to 27.75 MMOL/L | >27.76 MMOL/L or abnormal glucose with ketoacidosis or seizures |
| Hypocalcemia (corrected for albumin) | 2.10 to 1.95 MMOL/L | 1.94 to 1.75 MMOL/L | 1.74 to 1.52 MMOL/L | <1.52 MMOL/L or abnormal calcium with life-threatening arrhythmia or tetany |
| Hypercalcemia (corrected for albumin) | 2.64 to 2.87 MMOL/L | 2.88 to 3.12 | 3.13 to 3.37 MMOL/L | >3.37 MMOL/L or abnormal calcium with life-threatening arrhythmia |
| Hypomagnesemia | 0.7 to 0.6 MMOL/L | 0.59 to 0.45 MMOL/L | 0.44 to 0.3 MMOL/L | <0.3 MMOL/L or abnormal magnesium with life-threatening arrhythmia |
| Hypophosphatemia | 0.7 to 0.8 MMOL/L | 0.5 to 0.6 MMOL/L or replacement Rx required | 0.3 to 0.4 MMOL/L intensive therapy or hospitalization required | <0.3 MMOL/L or abnormal phosphate with life-threatening arrhythmia |
| Hyperbilirubinemia (when accompanied by any increase in other liver function test) | 1.1 to <1.25 × ULN | 1.25 to <1.5 × ULN | 1.5 to 1.75 × ULN | >1.75 × ULN |
| Hyperbilirubinemia (when other liver function tests are in the normal range) | 1.1 to <1.5 × ULN | 1.5 to <2.0 × ULN | 2.0 to 3.0 × ULN | >3.0 × ULN |
| Blood urea nitrogen | 1.25 to 2.5 × ULN | 2.6 to 5 × ULN | 5.1 to 10 × ULN | >10 × ULN |
| Hyperuricemia (uric acid) | 446 to 595 UMOL/L | 596 to 714 UMOL/L | 715 to 892 UMOL/L | >892 UMOL/L |
| Creatinine | 1.1 to 1.5 × ULN | 1.6 to 3.0 × ULN | 3.1 to 6.0 × ULN | >6 × ULN or dialysis required |

Rx = therapy; ULN = upper limit of normal.

| | Grade 1 | Grade 2 | Grade 3 | | Grade 4 |
|---|---|---|---|---|---|
| ENZYMES | | | | | |
| | | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Aspartate aminotransferase | | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alanine aminotransferase | | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Gamma to glutamyl transferase | | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alkaline Phosphatase | | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Amylase | | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |
| Lipase | | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |

ULN = upper limit of normal.

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Proteinuria | 1+ or | 2 to 3+ or | 4+ or | Nephrotic syndrome or |
| Fioleinuna | 200 MG to 1 GM loss/day | 1 to 2 GM loss/day | 2 to 3.5 GM loss/day | >3.5 GM loss/day |
| Hematuria | Microscopic only | Gross, no clots | Gross, with or without clots, | Obstructive or |
| пеннацина | <10 RBC/HPF | >10 RBC/HPF | or red blood cells casts | required transfusion |

HPF = high-powered field; RBC = red blood cells.

# 10.8. Appendix 8: Multiple Comparisons & Multiplicity

# 10.8.1. Handling of Multiple Comparisons & Multiplicity

No adjustments for multiplicity will be made.

# 10.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses.

# 10.9.1. Statistical Analysis Assumptions

| Endpoint(s) | <ul> <li>PK endpoints AUC(0-∞), AUC(0-t) and Cmax</li> </ul> |
|-------------|--------------------------------------------------------------|
| Analysis | Mixed Effects |

# **Assumptions:**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

# 10.10. Appendix 10 - Abbreviations & Trade Marks

# 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| Ae total | Total unchanged drug (total amount of drug excreted in urine) |
| Ae(t1-t2) | Amount of drug excreted in urine in a time interval |
| ANOVA | Analysis of variance |
| AUC(0-∞) | Area under the concentration-time curve from time zero (predose) |
| | extrapolated to infinite time |
| AUC(0-12) | Area under the urine concentration-time curve over time 0 (predose) to |
| | 12 hours after dosing. |
| AUC(0-24) | Area under the urine concentration-time curve over time 0 (predose) to |
| | 48 hours after dosing. |
| AUC(0-48) | Area under the urine concentration-time curve over time 0 (predose) to |
| | 48 hours after dosing. |
| AUC(0-t) | Area under the concentration-time curve from time zero (predose) to |
| | time of the last quantifiable concentration |
| BMI | Body mass index |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CLr | Renal clearance of drug |
| CV | Coefficient of variance |
| DNAUC(0-t) | Dose normalized area under the concentration-time curve from time 0 |
| 214100(01) | (predose) to time of the last quantifiable concentration |
| $DNAUC(0-\infty)$ | Dose normalized area under the concentration-time curve from time 0 |
| | (predose) extrapolated to infinite time |
| DNCmax | Dose normalized maximum observed concentration |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| fe% | Percentage of the given dose of drug excreted in urine |
| Frel | Relative bioavailability of drug |
| GSK | GlaxoSmithKline |
| hrs | Hours |
| HSWG | High shear wet granulation |
| IDSL | Integrated Data Standards Library |
| $\lambda z$ | Terminal phase rate constant |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligrams |
| msec | Milliseconds |
| %AUCex | The percentage of AUC (0-∞) obtained by extrapolation |
| PK | Pharmacokinetic |

| RAP | Reporting and Analysis Plan |
|------|----------------------------------------------------------------------|
| RC | Related compound |
| SAE | Serious Adverse Event(s) |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| t½ | Terminal half-life |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| Tmax | Time to first occurrence of Cmax |

# 10.10.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.11. Appendix 11: List of Data Displays

# 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|--------------|
| Study Population | 1.1 to 1.8 | |
| Safety | 2.1 to 2.12 | |
| Pharmacokinetic | 3.1 to 3.12 | 3.1 to 3.7.2 |
| Section | Listings | |
| ICH Listings | 1 to 44 | |

#### 10.11.2. Mock Example Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.11.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| IA [X] | Interim Analysis |
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.11.4. Study Population Tables

| Study Pop | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject D | isposition and | Analysis Sets | | | |
| 1.1 | Safety | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC [1] |
| 1.2 | Safety | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.3 | Screened | ES6 | Summary of Reasons for Screening Failures | | SAC [1] |
| 1.4 | Screened | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| Demograp | hics and Base | eline Characteris | stics | | |
| 1.5 | Safety | DM3 | Summary of Demographic Characteristics | | SAC [1] |
| 1.6 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |
| 1.7 | Safety | DM6 | Summary of Race and Racial Combinations Details | | SAC [1] |
| 1.8 | Safety | DM11 | Summary of Age Ranges | | SAC [1] |

# 10.11.5. Safety Tables

| Safety T | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Adverse | Events | | | | • |
| 2.1 | Safety | AE1 | Summary of All Adverse Events | | IA [1], SAC [1] |
| 2.2 | Safety | AE1 | Summary of All Drug- Related Adverse Events | | IA [1], SAC [1] |
| 2.3 | Safety | AE15 | Summary of Common (>=25%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | IA [1], SAC [1] |
| 2.4 | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | IA [1], SAC [1] |
| Laborat | ory Measureme | nts | | | • |
| 2.5 | Safety | LB1 | Summary of Clinical Chemistry Change from Baseline | | SAC [1] |
| 2.6 | Safety | LB1 | Summary of Haematology Change from Baseline | | SAC [1] |
| 2.7 | Safety | UR3b | Summary of Urinalysis Dipstick Results | | SAC [1] |
| Electro | cardiograms | | | | • |
| 2.8 | Safety | EG1 | Summary of ECG Findings | | SAC [1] |
| 2.9 | Safety | SAFE_T1 | Summary of Frequency of Maximum Post-Dose ECG Parameter Corrected QTc Interval | | SAC [1] |
| 2.10 | Safety | SAFE_T2 | Summary of Frequency of Maximum Change from Baseline for ECG Parameter Corrected QTc Interval | | SAC [1] |
| 2.11 | Safety | EG2 | Summary of Change from Baseline in ECG Values | | SAC [1] |
| Vital Sig | jns | | | | |
| 2.12 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC [1] |

# 10.11.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration Da | nta | | | |
| 3.1.1 | PK | PK01 | Summary of Plasma Gepotidacin Pharmacokinetic Concentration (ng/mL) - Time Data | | IA [1], SAC<br>[1] |
| 3.1.2 | PK | PK01 | Summary of Plasma Gepotidacin Pharmacokinetic Concentration (ng/mL) - Time Data – Excluding Outliers | exclude outliers | SAC [1] |
| 3.2 | PK | PK01 | Summary of Urine Gepotidacin Pharmacokinetic Concentration (ug/mL) - Time Data | | SAC [1] |
| PK Der | ived Paramete | ers | | | |
| 3.3.1 | PK | PKPT1 | Summary Statistics of Derived Plasma Gepotidacin Pharmacokinetic Parameters | Parameters with units | IA [1], SAC<br>[1] |
| 3.3.2 | PK | PKPT1 | Summary Statistics of Derived Plasma Gepotidacin<br>Pharmacokinetic Parameters – Excluding Outliers | Parameters with units, exclude outliers | SAC [1] |
| 3.3.3 | PK | PKPT1 | Summary Statistics of Pooled Derived Plasma<br>Gepotidacin Pharmacokinetic Parameters – Part 2<br>and 3 | Parameters with units | SAC [1] |
| 3.3.4 | PK | PKPT1 | Summary Statistics of Pooled Derived Plasma<br>Gepotidacin Pharmacokinetic Parameters – Part 2<br>and 3 Excluding Outliers | Parameters with units, exclude outliers | SAC [1] |
| 3.4 | PK | PKPT1 | Summary Statistics of Derived Urine Gepotidacin Pharmacokinetic Parameters | Parameters with units | SAC [1] |

| Pharm | acokinetic Tab | oles | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5.1 | PK | PKPT4 | Summary Statistics of Log-Transformed Derived Plasma Gepotidacin Pharmacokinetic Parameters | Parameters with units | IA [1], SAC<br>[1] |
| 3.5.2 | PK | PKPT4 | Summary Statistics of Log-Transformed Derived Plasma Gepotidacin Pharmacokinetic Parameters – Excluding Outliers | Parameters with units, exclude outliers | SAC [1] |
| 3.5.3 | PK | PKPT4 | Summary Statistics of Log-Transformed Pooled Derived Plasma Gepotidacin Pharmacokinetic Parameters – Part 2 and 3 | Parameters with units | SAC [1] |
| 3.5.4 | PK | PKPT4 | Summary Statistics of Log-Transformed Pooled Derived Plasma Gepotidacin Pharmacokinetic Parameters – Part 2 and 3 Excluding Outliers | Parameters with units, exclude outliers | SAC [1] |
| 3.6 | PK | PKPT4 | Summary Statistics of Log-Transformed Derived Urine Gepotidacin Pharmacokinetic Parameters | Parameters with units | SAC [1] |
| PK Ana | alysis Tables | | | | |
| 3.7 | PK<br>Parameter | PKPT3 | Analysis of Plasma Gepotidacin Pharmacokinetic Parameters by Treatment | AUC(0-t), AUC(0-∞), Cmax only log-transformed | IA [1], SAC<br>[1] |
| 3.8 | PK<br>Parameter | PK_T1 | Statistical Analysis of Plasma Gepotidacin Tmax by Treatment | Tmax Wilcox signed-rank test by group | IA [1], SAC<br>[1] |
| 3.9.1 | PK<br>Parameter | PKPT3 | Analysis of Dose-Normalized Plasma Gepotidacin<br>Pharmacokinetic Parameters for Fasted Japanese<br>Subjects | DNAUC(0-t), DNAUC(0-∞), DNCmax only log-<br>transformed by Treatment. Part 2 only. | SAC [1] |
| 3.9.2 | PK<br>Parameter | PKPT3 | Analysis of Dose-Normalized Plasma Gepotidacin<br>Pharmacokinetic Parameters for Fasted Japanese<br>Subjects – Excluding Outliers | DNAUC(0-t), DNAUC(0-∞), DNCmax only log-<br>transformed by Treatment. Part 2 only, exclude<br>outliers | SAC [1] |

| Pharmacokinetic Tables | | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title Programming Notes | | Deliverable<br>[Priority] | | |
| 3.9.3 | PK<br>Parameter | PKPT3 | Analysis of Dose-Normalized Plasma Gepotidacin<br>Pharmacokinetic Parameters for Pooled Japanese<br>Subjects | DNAUC(0-t), DNAUC(0-∞), DNCmax only log-<br>transformed by Treatment. Pooled Part 2 and 3<br>only | SAC [1] |
| 3.9.4 | PK<br>Parameter | PKPT3 | Analysis of Dose-Normalized Plasma Gepotidacin<br>Pharmacokinetic Parameters for Pooled Japanese<br>Subjects – Excluding Outliers | DNAUC(0-t), DNAUC(0-∞), DNCmax only log-<br>transformed by Treatment. Pooled Part 2 and 3<br>only, exclude outliers | SAC [1] |
| 3.10 | PK<br>Parameter | PKPT3 | Analysis of Dose Proportionality of Plasma<br>Gepotidacin Pharmacokinetic Parameters for Fed<br>Japanese Subjects | AUC(0-t), AUC(0-∞), Cmax only log-transformed by Treatment. Part 3 only. | SAC [1] |
| 3.11 | PK<br>Parameter | PK_T2 | Outliers Identified Using Grubbs' Test on Gepotidacin Plasma Pharmacokinetic Parameters | AUC(0-t), AUC(0-∞), Cmax | SAC [1] |

# 10.11.7. Pharmacokinetic Figures

| Pharma | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentra | tion Plots | | | |
| 3.1 | PK | PKCF1P | Individual Plasma Gepotidacin Concentration-Time Plots by Subject (Linear and Semi-Log) | Paginate by Subject | IA [1], SAC<br>[1] |
| 3.2 | PK | PKCF1P | Individual Urine Gepotidacin Concentration-Time Plots by Subject (Linear and Semi-Log) | Paginate by Subject | IA [1], SAC<br>[1] |
| Mean / | Median Conce | entration Plots | | | |
| 3.3.1 | PK | PKCF2 | Mean Plasma Gepotidacin Concentration-Time Plots by Treatment (Linear and Semi-log) | All treatments for each Part on one page | IA [1], SAC<br>[1] |
| 3.3.2 | PK | PKCF2 | Mean Plasma Gepotidacin Concentration-Time Plots by Treatment – Excluding Outliers (Linear and Semi-log) | All treatments for each Part on one page | SAC [1] |
| 3.4 | PK | PKCF2 | Mean Urine Gepotidacin Concentration-Time Plots by Treatment (Linear and Semi-log) | All treatments for each Part on one page | SAC [1] |
| 3.5.1 | PK | PKCF3 | Median Plasma Gepotidacin Concentration-Time Plots by Treatment (Linear and Semi-log) | All treatments for each Part on one page | IA [1], SAC<br>[1] |
| 3.5.2 | PK | PKCF3 | Median Plasma Gepotidacin Concentration-Time Plots by Treatment – Excluding Outliers (Linear and Semi-log) | All treatments for each Part on one page | SAC [1] |
| 3.6 | PK | PKCF3 | Median Urine Gepotidacin Concentration-Time Plots by Treatment (Linear and Semi-log) | All treatments for each Part on one page | SAC [1] |

| Pharma | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.7.1 | PK | PKPF3 | Individual and Box plot of Dose-Normalized Gepotidacin Plasma Pharmacokinetic Parameters by Treatment | Present PK parameters for each dose level Pages: Part 2 (2 doses) in one page, Part 3 (3 doses) in one page, and Part 2 and 3 in one page (Part 2 1500 mg, Part 3 1500 mg, Part 2 3000 mg, and Part 3 3000 mg) | SAC [1] |
| 3.7.2 | PK | PKPF3 | Individual and Box plot of Dose-Normalized Gepotidacin<br>Plasma Pharmacokinetic Parameters by Treatment –<br>Excluding Outliers | Present PK parameters for each dose level Pages: Part 2 (2 doses) in one page, Part 3 (3 doses) in one page, and Part 2 and 3 in one page (Part 2 1500 mg, Part 3 1500 mg, Part 2 3000 mg, and Part 3 3000 mg) | SAC [1] |
| 3.7.3 | PK | PKPF3 | Individual and Box plot of Pooled Dose-Normalized Gepotidacin Plasma Pharmacokinetic Parameters by Treatment – Part 2 and 3 | Present PK parameters for each dose level Pages: Pooled Part 2 and 3 DN parameters | SAC [1] |
| 3.7.4 | PK | PKPF3 | Individual and Box plot of Pooled Dose-Normalized<br>Gepotidacin Plasma Pharmacokinetic Parameters by<br>Treatment – Part 2 and 3 Excluding Outliers | Present PK parameters for each dose level Pages: Pooled Part 2 and 3 DN parameters | SAC [1] |

# 10.11.8. ICH Listings

| ICH : I | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | omisation | | | | |
| 1 | Safety | CP_TA1 | Listing of Randomised and Actual Treatment | | SAC [1] |
| Subje | ct Disposition | | | | |
| 2 | Safety | ES3 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC [1] |
| 4 | Screened | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 5 | Safety | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| 6 | Safety | SP3 | Listing of Subjects Excluded from Any Population | | SAC [1] |
| Demo | graphics | | | | |
| 7 | Safety | DM4 | Listing of Demographic Characteristics | Include height, weight and BMI | SAC [1] |
| 8 | Safety | DM10 | Listing of Race | | SAC [1] |
| Medic | al Conditions and | l Concomitant Medicat | ions | | |
| 9 | Safety | MH3 | Listing of Medical Conditions | | SAC [1] |
| 10 | Safety | CM4 | Listing of Concomitant Medications | | SAC [1] |
| Expos | sure | | | | |
| 11 | Safety | SAFE_L1 | Listing of Exposure Data | | SAC [1] |

| ICH: | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | 1 | | | | |
| 12 | Safety | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC[1] |
| 13 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [1] |
| 14 | Safety | SAFE_L2 | Listing of All Adverse Events | | IA[1], SAC [1] |
| 15 | Safety | AE9CP | Listing of Study Drug Related Adverse Events | | SAC [1] |
| 16 | Safety | AE9CP | Listing of Serious Adverse Events | | SAC [1] |
| 17 | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC [1] |
| 18 | Safety | SAFE_L3 | Listing of Liver Adverse Events | Conditional display | SAC [1] |
| 19 | Safety | SAFE_L4 | Listing of Cardiovascular Adverse Events | Conditional display | SAC [1] |
| 20 | Safety | SAFE_L5 | Listing of Allergic Reaction Adverse Events | Conditional display | SAC [1] |
| 21 | Safety | SAFE_L6 | Listing of Clostridium Difficile Testing | Conditional display | SAC [1] |
| 22 | Safety | SAFE_L7 | Listing of Rash Events | Conditional display | SAC [1] |
| Labor | atory Measureme | nts | | | |
| 23 | Safety | LB6 | Listing of Clinical Chemistry Toxicities of Grade 3 or Higher | | SAC [1] |
| 24 | Safety | LB6 | Listing of All Clinical Chemistry Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| 25 | Safety | LB6 | Listing of Haematology Toxicities of Grade 3 or Higher | | SAC [1] |
| 26 | Safety | LB6 | Listing of All Haematology Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| 27 | Safety | UR2b | Listing of Urinalysis Toxicities of Grade 3 or Higher | | SAC [1] |
| 28 | Safety | UR2b | Listing of All Urinalysis Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECGs | ECGs | | | | |
| 29 | Safety | EG6 | Listing of Abnormal ECG Findings | | SAC [1] |
| 30 | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC [1] |
| 31 | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance | | SAC [1] |
| 32 | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |
| 33 | Safety | SAFE_L8 | Listing of ECG Change from Baseline of Potential Clinical Importance | | SAC [1] |
| Vital S | Vital Signs | | | | |
| 34 | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance | | SAC [1] |
| 35 | Safety | VS5 | Listing of All Vital Signs for Subjects with Potential Clinical Importance Values | | SAC [1] |
| Liver | Events | | | | |
| 36 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Conditional display | SAC [1] |
| 37 | Safety | MH3 | Listing of Medical Conditions for Subjects with Liver Stopping Events | Conditional display | SAC [1] |
| 38 | Safety | SAFE_L10 | Listing of Alcohol Intake at Onset of Liver Event | Conditional display | SAC [1] |
| 39 | Safety | PKCL1X | Listing of Plasma Concentration Data for Subjects with Liver Stopping Events | Conditional display | SAC [1] |
| 40 | Safety | LIVER7 | Listing of Liver Biopsy Details | Conditional display | SAC [1] |
| 41 | Safety | LIVER8 | Listing of Liver Imaging Details | Conditional display | SAC [1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetic | | | | | |
| 42 | PK | PKCL1X | Listing of Plasma Gepotidacin Concentrations (ng/mL) by Treatment | Please list all the concentration data including unscheduled. Repeat for all treatments and Part 2 if needed. | SAC [1] |
| 43 | PK | PKCL1X | Listing of Urine Gepotidacin Concentrations (ug/mL) by Treatment | Please list all the concentration data including unscheduled. | SAC [1] |
| 44 | PK Parameter | PKPL1P | Listing of Gepotidacin Plasma Pharmacokinetic Parameters by Treatment | Additional parameters include Frel (units) (B and C only), t½ (units) and tlag (units). Repeat for Treatment B and C. Repeat for Treatments D and E if needed. | SAC [1] |

| ICH: | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 45 | PK Parameter | PKPL1P | Listing of Gepotidacin Urine Pharmacokinetic Parameters by Treatment | Additional parameters include Ae(0-2) (units), Ae(2-4) (units), Ae(4-6) units), Ae(8-12) (units), Ae(8-12) (units), Ae(12-24) (units), Ae(24-36) (units), Ae(36-48) (units), AUC(0-12) (units), AUC(0-24) (units), AUC(0-48) (units). Repeat for Treatments B and C. | SAC [1] |